CLINICAL TRIAL: NCT01254422
Title: Safety and Immunogenicity of a Tetravalent Dengue Vaccine in Healthy Children Aged 2 to 11 Years in Malaysia
Brief Title: Study of a Tetravalent Dengue Vaccine in Healthy Children Aged 2 to 11 Years in Malaysia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYD32; UTN: U1111-1115-6579 (Other: WHO)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue fever; Dengue hemorrhagic fever; CYD dengue vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue vaccine group (Experimental): Participants received 3 injections of the CYD dengue vaccine, 1 injection each at 0, 6, and 12 months.
  Interventions: Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus
- Placebo Group (Placebo Comparator): Participants received 3 injections of placebo, 1 injection each at 0, 6, and 12 months.
  Interventions: Biological: Placebo: NaCl 0.9%

INTERVENTIONS:
Biological: Live, attenuated, recombinant dengue serotypes 1, 2, 3, and 4 virus — 0.5 mL (at 0, 6, and 12 months), Subcutaneous suspension
  Other Names: CYD Dengue vaccine
  Arms: CYD Dengue vaccine group
Biological: Placebo: NaCl 0.9% — 0.5 mL (at 0, 6, and 12 months), Subcutaneous suspension
  Other Names: Saline
  Arms: Placebo Group

SUMMARY:
The purpose of this study was to evaluate the safety and immunogenicity of Phase III lots of the CYD dengue vaccine in a pediatric population in Malaysia.

Primary Objectives:

* To describe the safety (in terms of solicited and unsolicited adverse events) of the CYD dengue vaccine in all participants after each injection.
* To describe the antibody response to each dengue virus serotype post-injection 2 and post-injection 3.

DETAILED DESCRIPTION:
Healthy participants aged 2 to 11 years received 3 vaccinations at pre-determined schedules and were followed-up for at least 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 11 years on the day of inclusion
* Assent form was signed and dated by the participant (for participants ≥ 7 years) and informed consent form was signed and dated by the parent(s) or another legally accepted representative, and by an independent witness if the two parents or legally accepted representative were illiterate
* Participant and parent/legally accepted representative were able to attend all scheduled visits to comply with all trial procedures
* Participants in good health, based on medical history and physical examination
* For a female participant of childbearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to the first vaccination, until at least 4 weeks after the last vaccination

Exclusion Criteria:

* Known pregnancy, or a positive urine pregnancy test (for female participant of child-bearing potential only)
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Planned receipt of any vaccine in the 4 weeks following the trial first vaccination, except for pandemic influenza vaccination
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Seropositivity for human immunodeficiency virus (HIV) reported by the parent/legally acceptable representative
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion
* Participants who plan to move to another country/region within the 18 coming months
* Identified as a child (adopted or natural) of the Investigator or of site employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2012-09-28 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Singapore
Locations (4):
- Malaysia (4):
  - Ipoh, Perak
  - Kuala Lumpur
  - Kuching, Sarawak
  - Negeri Sembilan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Hss AS, Koh MT, Tan KK, Chan LG, Zhou L, Bouckenooghe A, Crevat D, Hutagalung Y. Safety and immunogenicity of a tetravalent dengue vaccine in healthy children aged 2-11 years in Malaysia: a randomized, placebo-controlled, Phase III study. Vaccine. 2013 Dec 2;31(49):5814-21. doi: 10.1016/j.vaccine.2013.10.013. Epub 2013 Oct 14. PMID 24135573
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 02 December 2010 to 10 February 2011 at 4 clinical sites in Malaysia.
Pre-assignment Details: A total of 250 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized.
Groups:
- CYD Dengue Vaccine Group: Participants received 3 injections (Inj.) of the CYD dengue vaccine, 1 injection each at 0, 6, and 12 months.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 199 | 51
Completed | 196 | 50
Not Completed | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Serious adverse event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants who were randomly assigned to CYD Dengue vaccine Group or Placebo Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 199 | 51 | 250
Age, Customized [Number; unit: Years]
  2 to 5 years | 99 | 26 | 125
  6 to 11 years | 100 | 25 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 19 | 122
  Male | 96 | 32 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Injection-site and Systemic Reactions Following Any and Each Vaccination With Either CYD Dengue Vaccine or a Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 Solicited injection site reactions: Pain: Incapacitating, unable to perform usual activities; Erythema and Swelling: >=50 millimeter (mm). Grade 3 Solicited systemic reactions: Fever: >=39°Degree Celsius (C); Headache, Malaise, Myalgia, and Asthenia: Significant: Prevents daily activity.
Time Frame: Day 0 up to Day 14 post-any and each vaccination
Population: Analysis was performed on safety analysis set which included participants who received any dose of CYD dengue vaccine or placebo and were analyzed according to the treatment received at this injection. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 199 | 51
Percentage of participants
  Inj. site Pain; Post-Any Inj. | 69.3 | 56.9
  Grade 3 Inj. site Pain; Post-Any Inj. | 1.0 | 0.0
  Inj. site Erythema; Post-Any Inj. | 46.7 | 49.0
  Grade 3 Inj. site Erythema; Post-Any Inj. | 0.5 | 0.0
  Inj. site Swelling; Post-Any Inj. | 38.7 | 35.3
  Grade 3 Inj. site Swelling; Post-Any Inj. | 0.5 | 0.0
  Inj. site Pain; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Inj. site Pain; Post-Inj. 1 | 41.4 | 27.5
  Grade 3 Inj. site Pain; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Grade 3 Inj. site Pain; Post-Inj. 1 | 0.5 | 0.0
  Inj. site Erythema; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Inj. site Erythema; Post-Inj. 1 | 22.2 | 23.5
  Grade 3 Inj. site Erythema; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Grade 3 Inj. site Erythema; Post-Inj. 1 | 0.5 | 0.0
  Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Inj. site Swelling; Post-Inj. 1 | 18.7 | 21.6
  Grade 3 Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Grade 3 Inj. site Swelling; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Inj. site Pain; Post-Inj. 2 | 48.2 | 26.0
  Grade 3 Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Inj. site Pain; Post-Inj. 2 | 0.5 | 0.0
  Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Inj. site Erythema; Post-Inj. 2 | 33.0 | 32.0
  Grade 3 Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Inj. site Erythema; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Inj. site Swelling; Post-Inj. 2 | 15.2 | 10.0
  Grade 3 Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Inj. site Swelling; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Inj. site Pain; Post-Inj. 3 | 40.0 | 38.0
  Grade 3 Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Inj. site Pain; Post-Inj. 3 | 0.5 | 0.0
  Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Inj. site Erythema; Post-Inj. 3 | 23.6 | 24.0
  Grade 3 Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Inj. site Erythema; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Inj. site Swelling; Post-Inj. 3 | 20.0 | 24.0
  Grade 3 Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Inj. site Swelling; Post-Inj. 3 | 0.5 | 0.0
  Asthenia; Post-Any Inj. | 47.2 | 33.3
  Grade 3 Asthenia; Post-Any Inj. | 3.0 | 0.0
  Fever; Post-Any Inj.: number analyzed (Participants) | 198 | 51
  Fever; Post-Any Inj. | 29.3 | 19.6
  Grade 3 Fever; Post-Any Inj.: number analyzed (Participants) | 198 | 51
  Grade 3 Fever; Post-Any Inj. | 6.6 | 3.9
  Headache; Post-Any Inj. | 52.3 | 39.2
  Grade 3 Headache; Post-Any Inj. | 2.0 | 2.0
  Malaise; Post-Any Inj. | 54.3 | 41.2
  Grade 3 Malaise; Post-Any Inj. | 3.5 | 0.0
  Myalgia; Post-Any Inj. | 37.7 | 31.4
  Grade 3 Myalgia; Post-Any Inj. | 2.5 | 0.0
  Asthenia; Post-Inj. 1 | 28.1 | 19.6
  Grade 3 Asthenia; Post-Inj. 1 | 2.0 | 0.0
  Fever; Post-Inj. 1: number analyzed (Participants) | 198 | 49
  Fever; Post-Inj. 1 | 12.6 | 8.2
  Grade 3 Fever; Post-Inj. 1: number analyzed (Participants) | 198 | 49
  Grade 3 Fever; Post-Inj. 1 | 2.0 | 4.1
  Headache; Post-Inj. 1 | 37.2 | 27.5
  Grade 3 Headache; Post-Inj. 1 | 1.5 | 0.0
  Malaise; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Malaise; Post-Inj. 1 | 36.4 | 29.4
  Grade 3 Malaise; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Grade 3 Malaise; Post-Inj. 1 | 2.5 | 0.0
  Myalgia; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Myalgia; Post-Inj. 1 | 22.7 | 23.5
  Grade 3 Myalgia; Post-Inj. 1: number analyzed (Participants) | 198 | 51
  Grade 3 Myalgia; Post-Inj. 1 | 2.0 | 0.0
  Asthenia; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Asthenia; Post-Inj. 2 | 23.9 | 6.0
  Grade 3 Asthenia; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Asthenia; Post-Inj. 2 | 0.5 | 0.0
  Fever; Post-Inj. 2: number analyzed (Participants) | 197 | 49
  Fever; Post-Inj. 2 | 15.2 | 10.2
  Grade 3 Fever; Post-Inj. 2: number analyzed (Participants) | 197 | 49
  Grade 3 Fever; Post-Inj. 2 | 2.5 | 0.0
  Headache; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Headache; Post-Inj. 2 | 31.0 | 16.0
  Grade 3 Headache; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Headache; Post-Inj. 2 | 0.5 | 2.0
  Malaise; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Malaise; Post-Inj. 2 | 27.9 | 6.0
  Grade 3 Malaise; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Malaise; Post-Inj. 2 | 0.5 | 0.0
  Myalgia; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Myalgia; Post-Inj. 2 | 18.8 | 8.0
  Grade 3 Myalgia; Post-Inj. 2: number analyzed (Participants) | 197 | 50
  Grade 3 Myalgia; Post-Inj. 2 | 0.5 | 0.0
  Asthenia; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Asthenia; Post-Inj. 3 | 19.0 | 12.0
  Grade 3 Asthenia; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Asthenia; Post-Inj. 3 | 1.5 | 0.0
  Fever; Post-Inj. 3: number analyzed (Participants) | 190 | 49
  Fever; Post-Inj. 3 | 9.5 | 2.0
  Grade 3 Fever; Post-Inj. 3: number analyzed (Participants) | 190 | 49
  Grade 3 Fever; Post-Inj. 3 | 3.7 | 0.0
  Headache; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Headache; Post-Inj. 3 | 22.6 | 14.0
  Grade 3 Headache; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Headache; Post-Inj. 3 | 1.5 | 0.0
  Malaise; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Malaise; Post-Inj. 3 | 20.5 | 12.0
  Grade 3 Malaise; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Malaise; Post-Inj. 3 | 1.5 | 0.0
  Myalgia; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Myalgia; Post-Inj. 3 | 17.4 | 10.0
  Grade 3 Myalgia; Post-Inj. 3: number analyzed (Participants) | 195 | 50
  Grade 3 Myalgia; Post-Inj. 3 | 1.0 | 0.0

2. Primary Outcome: Percentage of Flavivirus-Immune Participants Reporting Solicited Injection Site and Systemic Reactions Following Each Vaccination With CYD Dengue Vaccine or Placebo Vaccine
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Flavivirus-Immune participants were defined as participants with quantified antibodies against Japanese encephalitis and/or against at least 1 serotype with parental dengue virus strains (serotype 1, 2, 3, and 4) in the baseline sample.
Time Frame: Day 0 up to Day 14 post-each vaccination
Population: Analysis was performed on safety analysis set. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 111 | 31
Percentage of participants
  Injection site Pain; Post-Injection 1: number analyzed (Participants) | 110 | 31
  Injection site Pain; Post-Injection 1 | 44.5 | 29.0
  Injection site Erythema; Post-Injection 1: number analyzed (Participants) | 110 | 31
  Injection site Erythema; Post-Injection 1 | 14.5 | 29.0
  Injection site Swelling; Post-Injection 1: number analyzed (Participants) | 110 | 31
  Injection site Swelling; Post-Injection 1 | 13.6 | 22.6
  Asthenia; Post-Injection 1 | 27.9 | 25.8
  Fever; Post-Injection 1: number analyzed (Participants) | 110 | 30
  Fever; Post-Injection 1 | 12.7 | 13.3
  Malaise; Post-Injection 1: number analyzed (Participants) | 110 | 31
  Malaise; Post-Injection 1 | 38.2 | 38.7
  Myalgia; Post-Injection 1: number analyzed (Participants) | 110 | 31
  Myalgia; Post-Injection 1 | 22.7 | 25.8
  Headache; Post-Injection 1 | 36.9 | 29.0
  Injection site Pain; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Injection site Pain; Post-Injection 2 | 48.2 | 32.3
  Injection site Erythema; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Injection site Erythema; Post-Injection 2 | 25.5 | 29.0
  Injection site Swelling; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Injection site Swelling; Post-Injection 2 | 9.1 | 16.1
  Asthenia; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Asthenia; Post-Injection 2 | 21.8 | 9.7
  Fever; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Fever; Post-Injection 2 | 18.2 | 9.7
  Malaise; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Malaise; Post-Injection 2 | 29.1 | 3.2
  Myalgia; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Myalgia; Post-Injection 2 | 19.1 | 12.9
  Headache; Post-Injection 2: number analyzed (Participants) | 110 | 31
  Headache; Post-Injection 2 | 31.8 | 12.9
  Injection site Pain; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Injection site Pain; Post-Injection 3 | 34.3 | 41.9
  Injection site Erythema; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Injection site Erythema; Post-Injection 3 | 21.3 | 22.6
  Injection site Swelling; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Injection site Swelling; Post-Injection 3 | 15.7 | 22.6
  Asthenia; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Asthenia; Post-Injection 3 | 13.9 | 16.1
  Fever; Post-Injection 3: number analyzed (Participants) | 105 | 30
  Fever; Post-Injection 3 | 10.5 | 0.0
  Malaise; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Malaise; Post-Injection 3 | 18.5 | 16.1
  Myalgia; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Myalgia; Post-Injection 3 | 14.8 | 16.1
  Headache; Post-Injection 3: number analyzed (Participants) | 108 | 31
  Headache; Post-Injection 3 | 19.4 | 19.4

3. Primary Outcome: Percentage of Flavivirus-Naïve Participants Reporting Solicited Injection-site and Systemic Reactions Following Each Vaccination With CYD Dengue Vaccine or a Placebo Vaccine
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Flavivirus-Naive participants were defined as participants without quantified antibodies against Japanese encephalitis and without antibody quantified against all serotypes (1, 2, 3, and 4) with parental dengue virus strains in the baseline sample.
Time Frame: Day 0 up to Day 14 post-each vaccination
Population: Analysis was performed on safety analysis set. Here, ''overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 88 | 20
Percentage of participants
  Injection site Pain; Post-Injection 1 | 37.5 | 25.0
  Injection site Erythema; Post-Injection 1 | 31.8 | 15.0
  Injection site Swelling; Post-Injection 1 | 25.0 | 20.0
  Asthenia; Post-Injection 1 | 28.4 | 10.0
  Fever; Post-Injection 1: number analyzed (Participants) | 88 | 19
  Fever; Post-Injection 1 | 12.5 | 0.0
  Malaise; Post-Injection 1 | 34.1 | 15.0
  Myalgia; Post-Injection 1 | 22.7 | 20.0
  Headache; Post-Injection 1 | 37.5 | 25.0
  Injection site Pain; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Injection site Pain; Post-Injection 2 | 48.3 | 15.8
  Injection site Erythema; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Injection site Erythema; Post-Injection 2 | 42.5 | 36.8
  Injection site Swelling; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Injection site Swelling; Post-Injection 2 | 23.0 | 0.0
  Asthenia; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Asthenia; Post-Injection 2 | 26.4 | 0.0
  Fever; Post-Injection 2: number analyzed (Participants) | 87 | 18
  Fever; Post-Injection 2 | 11.5 | 11.1
  Malaise; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Malaise; Post-Injection 2 | 26.4 | 10.5
  Myalgia; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Myalgia; Post-Injection 2 | 18.4 | 0.0
  Headache; Post-Injection 2: number analyzed (Participants) | 87 | 19
  Headache; Post-Injection 2 | 29.9 | 21.1
  Injection site Pain; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Injection site Pain; Post-Injection 3 | 47.1 | 31.6
  Injection site Erythema; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Injection site Erythema; Post-Injection 3 | 26.4 | 26.3
  Injection site Swelling; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Injection site Swelling; Post-Injection 3 | 25.3 | 26.3
  Asthenia; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Asthenia; Post-Injection 3 | 25.3 | 5.3
  Fever; Post-Injection 3: number analyzed (Participants) | 85 | 19
  Fever; Post-Injection 3 | 8.2 | 5.3
  Malaise; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Malaise; Post-Injection 3 | 23.0 | 5.3
  Myalgia; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Myalgia; Post-Injection 3 | 20.7 | 0.0
  Headache; Post-Injection 3: number analyzed (Participants) | 87 | 19
  Headache; Post-Injection 3 | 26.4 | 5.3

4. Primary Outcome: Percentage of Participants With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Seropositivity was defined as participants achieving neutralizing antibody titers >=10 (1/dilution) against each dengue serotype (1,2, 3 and 4) and was assessed using the Dengue Plaque Reduction Neutralization Test (PRNT).
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set which included participants who received at least one injection of CYD dengue vaccine or placebo and had at least one valid post-injection serology result. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 196 | 50
Percentage of participants
  Serotype 1; Pre-Injection 1 | 31.1 | 32.0
  Serotype 1; Post-Injection 2 | 90.3 | 34.0
  Serotype 1; Post-Injection 3 | 96.4 | 30.0
  Serotype 2; Pre-Injection 1 | 27.6 | 30.0
  Serotype 2; Post-Injection 2 | 94.9 | 34.0
  Serotype 2; Post-Injection 3 | 96.9 | 34.0
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 196 | 49
  Serotype 3; Pre-Injection 1 | 36.7 | 36.7
  Serotype 3; Post-Injection 2 | 98.5 | 32.0
  Serotype 3; Post-Injection 3 | 99.0 | 34.0
  Serotype 4; Pre-Injection 1 | 24.0 | 30.0
  Serotype 4; Post-Injection 2 | 91.8 | 32.0
  Serotype 4; Post-Injection 3 | 98.0 | 28.0

5. Primary Outcome: Percentage of Participants With Seropositivity Against at Least One, Two, Three, or the Four Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: Seropositivity was defined as participants achieving neutralizing antibody titers >=10 (1/dilution) against each dengue serotype (1, 2, 3, and 4) and was assessed using the dengue PRNT.
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 196 | 50
Percentage of participants
  At least 1 serotype; Pre-Injection 1 | 44.9 | 48.0
  At least 1 serotype; Post-Injection 2 | 100.0 | 46.0
  At least 1 serotype; Post-Injection 3 | 100.0 | 42.0
  At least 2 serotypes; Pre-Injection 1 | 29.1 | 28.0
  At least 2 serotypes; Post-Injection 2 | 99.0 | 34.0
  At least 2 serotypes; Post-Injection 3 | 100.0 | 32.0
  At least 3 serotypes; Pre-Injection 1 | 25.5 | 28.0
  At least 3 serotypes; Post-Injection 2 | 96.4 | 28.0
  At least 3 serotypes; Post-Injection 3 | 98.5 | 30.0
  All 4 serotypes; Pre-Injection 1 | 19.9 | 24.0
  All 4 serotypes; Post-Injection 2 | 80.1 | 24.0
  All 4 serotypes; Post-Injection 3 | 91.8 | 22.0

6. Primary Outcome: Geometric Mean Titers (GMTs) Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: GMTs of antibodies against the dengue virus serotypes (1, 2, 3, and 4) were assessed using the dengue PRNT.
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 196 | 50
Titers (1/dilution)
  Serotype 1; Pre-Injection 1 | 15.3 [11.5 to 20.4] | 18.6 [9.69 to 35.8]
  Serotype 1; Post-Injection 2 | 119 [90.7 to 155] | 21.0 [10.6 to 41.9]
  Serotype 1; Post-Injection 3 | 151 [121 to 188] | 18.9 [9.94 to 35.8]
  Serotype 2; Pre-Injection 1 | 15.9 [11.8 to 21.3] | 18.6 [10.0 to 34.5]
  Serotype 2; Post-Injection 2 | 160 [127 to 203] | 17.9 [9.91 to 32.2]
  Serotype 2; Post-Injection 3 | 180 [146 to 221] | 16.3 [9.59 to 27.7]
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 196 | 49
  Serotype 3; Pre-Injection 1 | 15.6 [12.3 to 19.9] | 15.9 [9.57 to 26.5]
  Serotype 3; Post-Injection 2 | 196 [163 to 235] | 15.9 [9.27 to 27.4]
  Serotype 3; Post-Injection 3 | 193 [161 to 231] | 16.3 [9.81 to 27.0]
  Serotype 4; Pre-Injection 1 | 9.92 [8.17 to 12.0] | 12.3 [7.96 to 19.0]
  Serotype 4; Post-Injection 2 | 110 [88.9 to 136] | 13.3 [7.94 to 22.1]
  Serotype 4; Post-Injection 3 | 114 [97.0 to 134] | 10.9 [7.34 to 16.2]

7. Primary Outcome: Percentage of Participants With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo: Flavivirus-Immune Participants
Description: Seropositivity was defined as participants achieving neutralizing antibody titers >=10 (1/dilution) against each serotype (1, 2, 3, and 4) and was assessed using the Dengue PRNT. Flavivirus-Immune participants were defined as participants with quantified antibodies against Japanese encephalitis and/or against at least 1 serotype (1, 2, 3, and 4) with parental dengue virus strains in the baseline sample.
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: Analysis was performed on Full analysis set. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 109 | 31
Percentage of participants
  Serotype 1; Pre-Injection 1 | 56.0 | 51.6
  Serotype 1; Post-Injection 2 | 96.3 | 48.4
  Serotype 1; Post-Injection 3 | 97.2 | 41.9
  Serotype 2; Pre-Injection 1 | 49.5 | 48.4
  Serotype 2; Post-Injection 2 | 96.3 | 54.8
  Serotype 2; Post-Injection 3 | 97.2 | 48.4
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 109 | 30
  Serotype 3; Pre-Injection 1 | 66.1 | 60.0
  Serotype 3; Post-Injection 2 | 100.0 | 51.6
  Serotype 3; Post-Injection 3 | 99.1 | 48.4
  Serotype 4; Pre-Injection 1 | 43.1 | 48.4
  Serotype 4; Post-Injection 2 | 97.2 | 45.2
  Serotype 4; Post-Injection 3 | 100.0 | 41.9

8. Primary Outcome: Percentage of Participants With Seropositivity Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo: Flavivirus-Naive Participants
Description: Seropositivity was defined as participants achieving neutralizing antibody titers >=10 (1/dilution) against each serotype (1, 2, 3, and 4) and was assessed using the Dengue PRNT. Flavivirus naïve participants were defined as participants without quantified antibodies against Japanese encephalitis and without quantified antibodies against all serotypes (1, 2, 3, and 4) with parental dengue virus strains in the baseline sample.
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 87 | 19
Percentage of participants
  Serotype 1; Pre-Injection 1 | 0.0 | 0.0
  Serotype 1; Post-Injection 2 | 82.8 | 10.5
  Serotype 1; Post-Injection 3 | 95.4 | 10.5
  Serotype 2; Pre-Injection 1 | 0.0 | 0.0
  Serotype 2; Post-Injection 2 | 93.1 | 0.0
  Serotype 2; Post-Injection 3 | 96.6 | 10.5
  Serotype 3; Pre-Injection 1 | 0.0 | 0.0
  Serotype 3; Post-Injection 2 | 96.6 | 0.0
  Serotype 3; Post-Injection 3 | 98.9 | 10.5
  Serotype 4; Pre-Injection 1 | 0.0 | 0.0
  Serotype 4; Post-Injection 2 | 85.1 | 10.5
  Serotype 4; Post-Injection 3 | 95.4 | 5.3

9. Primary Outcome: GMTs of Flavivirus-Immune Participants Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: GMTs of antibodies against the dengue virus serotypes (1, 2, 3, and 4) were assessed using the Dengue PRNT. Flavivirus-Immune participants were defined as participants with quantified antibodies against Japanese encephalitis and/or against at least 1 serotype (1, 2, 3, and 4) with parental dengue virus strains in the baseline sample.
Time Frame: Pre-Injection 1 and Post-Injections 2 and 3
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 109 | 31
Titers (1/dilution)
  Serotype 1; Pre-Injection 1 | 37.5 [24.0 to 58.6] | 41.7 [16.0 to 109]
  Serotype 1; Post-Injection 2 | 248 [171 to 361] | 45.4 [16.3 to 127]
  Serotype 1; Post-Injection 3 | 247 [178 to 343] | 33.5 [13.3 to 84.4]
  Serotype 2; Pre-Injection 1 | 39.9 [25.2 to 63.1] | 41.6 [17.0 to 102]
  Serotype 2; Post-Injection 2 | 306 [221 to 424] | 39.0 [16.7 to 91.3]
  Serotype 2; Post-Injection 3 | 292 [217 to 395] | 30.0 [13.8 to 64.9]
  Serotype 3; Pre-Injection 1: number analyzed (Participants) | 109 | 30
  Serotype 3; Pre-Injection 1 | 38.8 [27.3 to 55.4] | 33.2 [16.1 to 68.5]
  Serotype 3; Post-Injection 2 | 296 [230 to 381] | 32.4 [14.8 to 71.0]
  Serotype 3; Post-Injection 3 | 287 [219 to 376] | 29.5 [14.2 to 61.1]
  Serotype 4; Pre-Injection 1 | 17.1 [12.5 to 23.5] | 21.3 [11.3 to 40.1]
  Serotype 4; Post-Injection 2 | 152 [115 to 201] | 21.7 [10.0 to 46.9]
  Serotype 4; Post-Injection 3 | 155 [125 to 191] | 16.5 [9.17 to 29.7]

10. Primary Outcome: GMT of Flavivirus-Naïve Participants Against Each Serotype With the Parental Dengue Virus Strains Before and After Vaccinations With Either CYD Dengue Vaccine or a Placebo
Description: GMTs of antibodies against the dengue virus serotypes (1, 2, 3, and 4) were assessed using the Dengue PRNT. Flavivirus-Naive participants were defined as participants without quantified antibodies against Japanese encephalitis and without antibody quantified against all serotypes (1, 2, 3, and 4) with parental dengue virus strains in the baseline sample.
Time Frame: Pre-Injection 1 and Post- Injections 2 and 3
Population: Analysis was performed on Full analysis set. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 87 | 19
Titers (1/dilution)
  Serotype 1; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 1; Post-Injection 2 | 47.1 [35.3 to 62.9] | 5.98 [4.62 to 7.74]
  Serotype 1; Post-Injection 3 | 81.6 [66.3 to 101] | 7.38 [3.88 to 14.0]
  Serotype 2; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-Injection 2 | 71.4 [55.4 to 92.1] | 5.00 [5.00 to 5.00]
  Serotype 2; Post-Injection 3 | 97.5 [77.5 to 123] | 6.03 [4.43 to 8.21]
  Serotype 3; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-Injection 2 | 116 [92.6 to 146] | 5.00 [5.00 to 5.00]
  Serotype 3; Post-Injection 3 | 117 [97.4 to 141] | 6.17 [4.52 to 8.41]
  Serotype 4; Pre-Injection 1 | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  Serotype 4; Post-Injection 2 | 73.3 [53.7 to 100] | 5.95 [4.47 to 7.91]
  Serotype 4; Post-Injection 3 | 78.0 [62.0 to 98.1] | 5.54 [4.47 to 6.87]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Day 0 (post-vaccination) up to 6 months post-Injection 3 (up to 18 months)
Description: Analysis was performed on Safety analysis set.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/51
Serious Adverse Events (participants affected / at risk) | 11/199 | 7/51
Other Adverse Events (participants affected / at risk) | 138/199 | 29/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=199) | Placebo Group (N=51)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=199) | Placebo Group (N=51)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 1 (1)
Headache; Post-Any Injection (Nervous system disorders) | 104 (104) | 20 (20)
Pyrexia (General disorders) | 14 (14) | 1 (1)
Injection site Pain; Post-Any (General disorders) | 138 (138) | 29 (29)
Injection site Erythema; Post-Any (General disorders) | 93 (93) | 25 (25)
Injection site Swelling; Post-Any (General disorders) | 77 (77) | 18 (18)
Asthenia; Post-Any Injection (General disorders) | 94 (94) | 17 (17)
Fever; Post-Any Injection (General disorders) | 58/198 (58) | 10 (10)
Malaise; Post-Any Injection (General disorders) | 108 (108) | 21 (21)
Vomiting (Gastrointestinal disorders) | 7 (7) | 3 (3)
Myalgia; Post-Any Injection (Musculoskeletal and connective tissue disorders) | 75 (75) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 50 (61) | 11 (15)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.